CLINICAL TRIAL: NCT01373047
Title: Phase I Trial Of Intrahepatic Infusion Of 2nd Generation Designer T Cells For Cea-Expressing Liver Metastases
Brief Title: CEA-Expressing Liver Metastases Safety Study of Intrahepatic Infusions of Anti-CEA Designer T Cells
Acronym: HITM
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Roger Williams Medical Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RWH 335-99
Record Dates: First submitted 2011-06-09; First posted 2011-06-14 (Estimated); Last update posted 2013-07-30 (Estimated); Status verified 2013-07

CONDITIONS: Liver Metastases
Keywords: liver metastases; immunotherapy; regional therapy; T cells

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Intrahepatic anti-CEA designer T cells (Experimental)
  Interventions: Biological: anti-CEA 2nd generation designer T cells

INTERVENTIONS:
Biological: anti-CEA 2nd generation designer T cells — Three infusions of gene-modified T cells over the course of 6 weeks into the hepatic artery via a percutaneous approach.
  Other Names: anti-CEA T cells; designer T cells

SUMMARY:
The purpose of this study is to collect data on the safety and potential effectiveness of 2nd generation designer T cells delivered into the hepatic circulation in patients with liver metastases expressing the CEA tumor marker. Designer T cells are prepared by collecting white blood cells from the participant, and then modifying these cells in the laboratory so that they recognize the tumor antigen, CEA. These modified cells are then given back into the participant so that they can attack and kill tumor cells. The investigators hypothesize that regional delivery of the designer T cells directly into the hepatic artery will minimize systemic toxicity and optimize the changes for therapeutic effect.

DETAILED DESCRIPTION:
T cells have the power to destroy malignant cells under certain conditions, as demonstrated by the rare spontaneous remissions of cancer. However, the endogenous T cell response to cancer fails in the vast majority of patients and the tolerogenic conditions within the liver may pose additional immunologic barriers for those with intrahepatic metastases. The investigators modify patient T cells to kill malignant cells based on their expression of tumor antigens using antibody-defined recognition. The investigators will achieve this by preparing chimeric IgCD28TCR genes in mammalian expression vectors to yield "designer T cells" from normal patient cells. Prior studies in model systems demonstrated that recombinant IgCD28TCR could direct modified T cells to respond to antigen targets with IL2 secretion, cellular proliferation, and cytotoxicity - the hallmarks of an effective, self-sustaining immune response.

The present trial will test the regional infusion of anti-CEA designer T cells, given via the hepatic artery using a percutaneous approach. This is an intra-patient dose escalation trial, where patients will receive three doses over the course of six weeks. Doses are 10^8, 10^9 and 10^10 modified T cells. Patients are monitored for safety and response. Patients are on-study for one month after dosing.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed diagnosis of CEA+ adenocarcinoma and liver metastases
* Liver metastases must be CEA-expressing as demonstrated by elevated serum CEA levels (≥10ng/ml) or immunohistochemistry on a biopsy specimen
* Failure on at least one line of standard systemic chemotherapy and have unresectable liver disease
* Measurable liver disease (> 1.0 cm by CT or MRI)
* Extrahepatic disease is acceptable when limited to the lungs and/or abdominal lymph nodes
* At least 18 years of age
* Able to understand and sign informed consent
* Life expectancy of greater than four months
* Good performance status (PS 0-1)

Exclusion Criteria:

* Pregnancy
* Serious medical conditions including but not limited to liver, cardiopulmonary, and renal disease
* Patients with a history of portal hypertension, cirrhosis, hepatitis, or with radiographic evidence of cirrhosis
* Concurrent malignancy
* Use of systemic steroids

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2011-06; Primary Completion 2013-07 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
Determine the safety of modified T cells delivered into the hepatic artery by documenting the type and severity of any side effects and establishing the Maximum Tolerated Dose (MTD). | 1 month

SECONDARY OUTCOMES:
Tumor Response by CT or MRI and PET scan | 1 month
  CT or MRI and PET imaging will be obtained before the first infusion and following the final infusion to document changes in liver tumor size and metabolic activity.
Designer T cell distribution following infusion | 1 month
  Using liver tumor biopsy specimens and blood collection, we will determine the extent to which infused T cells enter the liver tumors in addition to circulation in the extrahepatic space.
Designer T cell survival and phenotype following infusion | 1 month
  Using tissue obtained from biopsies in addition to blood samples, the duration of T cell persistence will be assessed, in addition to cell surface markers.

CONTACTS AND LOCATIONS:
Overall Officials: Steven C Katz, MD, Principal Investigator — Roger Williams Medical Center
Locations (1):
- Roger Williams Medical Center, Providence, Rhode Island, United States

REFERENCES:
- See also: Roger Williams Surgical Oncology — http://www.rhodeislandcancer.org